CLINICAL TRIAL: NCT03919812
Title: Immunomodulatory Effect of Vitamin D Supplementation on Monocyte in Major Beta-thalassemia
Brief Title: Immunomodulatory Vitamin D in Thalassemia
Acronym: ThalTB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Collaborators: Hasan Sadikin General Hospital (Other)
Responsible Party: Principal Investigator, Mohammad Ghozali, Principal Investigator, Universitas Padjadjaran
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TB-201804.01
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Thalassemia; Tuberculosis; Vitamin D Deficiency
MeSH Terms: conditions — Thalassemia; Tuberculosis; Vitamin D Deficiency

STUDY DESIGN:
Intervention Model Description: This study was designed as a non-randomized, open label, intervention study and performed at the thalassemia clinic of the Hasan Sadikin General Hospital, Bandung, West Java, Indonesia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitamin D supplementation according to baseline Vitamin D (Experimental): The intervention provided according to the participants' state of vitamin D sufficiency. vitamin D sufficient participants received 800 IU cholecalciferol (syrup containing 400 IU cholecalciferol per measuring spoon, Gracia Pharmindo, Indonesia) daily for 8 weeks, while those who had insufficient or deficient vitamin D level consumed 2000 IU daily. Compliance was systematically monitored using drug monitoring diary evaluated by researchers. Blood samples for the study objectives were taken at enrollment and after eight weeks of cholecalciferol supplementation during routinely scheduled visits to the clinic.
  Interventions: Dietary Supplement: Cholecalciferol supplementation

INTERVENTIONS:
Dietary Supplement: Cholecalciferol supplementation — supplementation received by subject according to their vitamin D status: insufficiency or deficiency.

SUMMARY:
Thalassemia becomes one of global health issue and so does Indonesia. In 2015, more than 7600 children were diagnosed as this hemoglobin genetic disease wherein anemia and lifetime blood transfusion contribute to their morbidity and mortality in Indonesia. Major β-Thalassemia is the most common type found. However, along with disease progression and age, iron accumulation and dysregulation becomes the most common complication exist. In cellular level, this condition results in cell and tissue damage especially immune cells and promotes favor condition for siderophilic bacteria such as Mycobaterium tuberculosis (Mtb) to growth rapidly. Severe infection becomes the second most cause of death in thalassemia-β major patients.

Tuberculosis (Tb) remains the global health issue especially in developing countries. Based on World Health Organization (WHO) report on 2015, Indonesia is the second highest burden of TB in the world. Both of adaptive and innate immune system plays important role in Mtb recognition and eradication. However, immune cells mechanism and activity in response to Mtb infection during iron accumulation condition on thalassemia-β major patients may be altered therefore need for further study. Macrophage is an adaptive immune cell, has a pivotal role on circulating-iron regulation and serves as Mtb host cell. To understand macrophage activity on thalassemia-β major patients can be studied by monocyte characteristic stimulated by Mtb antigen and evaluated by its differentiation into three subsets based on CD14 and CD16. Mtb antigen presentation is identified by HLA-DR expression on monocyte membrane.

Vitamin D is one of the most affected micronutrients on major β-thalassemia patients, yet it has immunomodulatory effect on immune system. Recent finding of vitamin D receptor (VDR) expressed in monocyte strongly convince that vitamin D should be maintained in major β-thalassemia patients where it is found lower in these patients. Thus, this original and true report aimed to declare that the research activity has finished and the data has been elaborated. Future plan is developing the original article based on the research finding corroborating the previous knowledge and innovative suggestion for the quality of thalassemia.

DETAILED DESCRIPTION:
This study was designed as a non-randomized, open label, intervention study and performed at the thalassemia clinic of the Hasan Sadikin General Hospital, Bandung, West Java, Indonesia. Vitamin D deficiency in the general population is common in Indonesia with a prevalence of 41% reported in one study1. Sixty children (aged 1 month to 15 years) diagnosed as major β-thalassemia confirmed by clinical and hemoglobin electrophoresis who regularly having blood transfusion at least once in a month controlled in the clinic, from March - May 2018 were recruited prospectively. In addition, children who had ferritin serum >1000 µg/L in the last three months were met criteria for enrollment. Children who had tuberculosis or co-infection (hepatitis B, hepatitis C, and cytomegalovirus) and sign of acute infection were not eligible for enrollment. Informed consent was obtained from parents or child's guardian. Vitamin D levels were measured before and after supplementation while identifying their vitamin D sufficiency status. Classification of vitamin D sufficiency were used according to The Endocrine Society Clinical Practice Guideline, which stated that the level of 25(OH)D of < 20 ng/ml was considered to be vitamin D deficiency whereas a 25(OH)D of 21-29 ng/ml was considered to be insufficient. Then, a sufficient vitamin D was considered when the concentration of 25(OH)D was 30 ng/mL or above.2 No healthy control was enrolled to test for variability in the laboratory tests over time in this study.

The intervention provided according to the participants' state of vitamin D sufficiency. vitamin D sufficient participants received 800 IU cholecalciferol (syrup containing 400 IU cholecalciferol per measuring spoon, Gracia Pharmindo, Indonesia) daily for 8 weeks, while those who had insufficient or deficient vitamin D level consumed 2000 IU daily. Compliance was systematically monitored using drug monitoring diary evaluated by researchers. Blood samples for the study objectives were taken at enrollment and after eight weeks of cholecalciferol supplementation during routinely scheduled visits to the clinic. The outcome measure was the change in the proportion of monocyte subsets and the expression of membrane-bound protein of monocyte consist of CD14, CD16, and HLA-DR.

All procedures were conducted in accordance with policies of the Faculty of Medicine, Universitas Padjadjaran and Hasan Sadikin General Hospital, Bandung, West Java, Indonesia. This study was approved by Health Research Ethics Committee of Medical Faculty Universitas Padjadjaran Bandung with approval number 50/UN6.KEP/EC/2018. All participants signed a written informed consent. All participants signed a written informed consent. This study was registered in clinicaltrial.gov

ELIGIBILITY:
Inclusion Criteria:

* Children (aged 1 month to 15 years) diagnosed as major β-thalassemia
* Regularly having blood transfusion at least once in a month
* controlled in Thalassemia Polyclinic of Hasan Sadikin General Hospital Bandung, West Java,
* had ferritin serum >1000 µg/L in the last three months

Exclusion Criteria:

* Children who had co-infection (hepatitis B, hepatitis C, and cytomegalovirus) and sign of acute infection were not eligible for enrollment.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
The outcome measure was the change in the proportion of monocyte subsets | Eight-week supplementation
  The outcome measure was the change in the proportion of monocyte subsets and the expression of membrane-bound protein of monocyte consist of CD14, CD16, and HLA-DR.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Ghozali, Dr., Principal Investigator — Faculty of Medicine Universitas Padjadjaran
Locations (1):
- Klinik Thalassemia Rumah Sakit Dr. Hasan Sadikin Bandung, Bandung, West Java, Indonesia